CLINICAL TRIAL: NCT02667249
Title: Compliance of Clinical Pathways in Elective Laparoscopic Cholecystectomy: Evaluation of Different Implementation Methods
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: ICP 001
Record Dates: First submitted 2015-12-08; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2015-11

CONDITIONS: Gallstones
Keywords: cholecystectomy, check list
MeSH Terms: conditions — Gallstones | interventions — Critical Pathways

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- check list: clinical pathway using a paper based check-list
  Interventions: Other: clinical pathway
- integrated clinical pathway: clinical pathway in form of a clinical pathway integrated into the paper based medical treatment and nursing documentation
  Interventions: Other: clinical pathway

INTERVENTIONS:
Other: clinical pathway — implementation of a standardized clinical pathway

SUMMARY:
Compliance to the clinical pathway, postoperative complication and total cost of the hospitalisation of patients undergoing elective cholecystectomy for symptomatic cholecystolithiasis were collected over two different periods: using a clinical pathway in form of a paper based check-list (group 1, n=118) or a clinical pathway integrated into the paper based medical treatment and nursing documentation (group 2, n=123). Outcome measures were compliance of the clinical pathway and total costs per case.

DETAILED DESCRIPTION:
Data of patients undergoing elective cholecystectomy for symptomatic cholecystolithiasis were collected over two different periods: a clinical pathway in form of a paper based check-list (check-list group, n=118, or in form of a clinical pathway integrated into the paper based medical treatment and nursing documentation (integrated clinical pathway group, n=123. A standardized clinical pathway for elective laparoscopic cholecystectomy in form of a check list was initially established in 2008 and evaluated during a 6-month period (August 2011 until January 2012) at the University of Tuebingen. The integrated clinical pathway was evaluated during a 6-month period after an introduction phase of 2 months (November 2012 until April 2013). The contents of both clinical pathways were identical, especially concerning the standardization of perioperative fluid management, perioperative monitoring, nutrition, analgesia, reserve medications, preoperative and postoperative examinations, detailed laboratory blood testing, nursing standards and planned discharge.

Primary outcome measure was the compliance to the clinical pathway defined as an adherence of more than 80% to the presetted pathway items.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective laparoscopic cholecystectomy

Exclusion Criteria:

* emergency procedures
* conversion to open cholecystectomy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective laparoscopic cholecystectomy
Sampling Method: Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2011-08; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
compliance to clinical pathway | time period which is covered by the clinical pathway beginning from preclinical check up until final discharge after cholecystctomy (usually a time frame of 7-14 days)
  Compliance to clinical pathway defined as an adherence of more than 80% to the presetted pathway items as reported on a paper based check-list

SECONDARY OUTCOMES:
complication | 30 days complication rate
  Complications assessed according to Clavien classification 30 days postoperative
total cost | total cost of the hospitalization covering the period from preclinical check up until final discharge after cholecystctomy (usually a time frame of 7-14 days)
  total costs per case covering the period from preclinical check up until final and discharge after cholecystctomy (€) were assessed using our prospective. electronic patient and quality assessment data base. Costs were calculated according to our internal transfer prices.

IPD SHARING:
Plan to Share IPD: No